CLINICAL TRIAL: NCT05656222
Title: A Retrospective Study Investigating the Combination of Irinotecan, Vincristine and Anlotinib for Epithelioid Sarcoma
Brief Title: Irinotecan and Anlotinib for Epithelioid Sarcoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Check the IRB again
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xie Lu, Musculoskeletal Tumor Center, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-sarcoma 15
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Objective Response; Overall Survival
Keywords: Epithelioid sarcoma; systemic treatment; objective response; toxicity
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VIA treatment Group (Experimental)
  Interventions: Drug: VIA combination treatment

INTERVENTIONS:
Drug: VIA combination treatment — a 90-minute intravenous infusion of irinotecan at a dose of 50 mg/m2/d for 5 days every 3 weeks, vincristine given at a dose of 1.4 mg/m2 (maximum 2 mg) on days 1 and 8, and oral administration of Anlotinib once daily on days 1-14 within a 21-day cycle.

SUMMARY:
Epithelioid sarcoma is a rare soft tissue sarcoma characterized by SMARCB1/INI1 deficiency. Much attention has been paid to the selective EZH2 inhibitor tazemetostat, where other systemic treatments are generally ignored. To explore alternative treatment options, we studied the effects of irinotecan-based chemotherapy in a series of epithelioid sarcoma patients.

ELIGIBILITY:
Inclusion Criteria:

* (1) Grade 2 or 3 ES confirmed histologically using the American Joint Committee on Cancer (AJCC) system ;
* (2) patients presented with measurable lesions using the Response Evaluation Criteria In Solid Tumors (RECIST1.1) and were not amenable to surgical resection or radiotherapy;
* (3) primary or secondary metastatic disease;
* (4) received more than two courses of the VIA regimen;
* (5) no concurrent treatment was given while on the VIA regimen;
* (6) follow-up information and evaluation after chemotherapy were available.

Exclusion Criteria:

* less than 4 cycles of treatment;
* medical records were not complete.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 12 weeks
  Based on RECIST1.1 criteria, clinical evaluation was done once every 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

REFERENCES:
- [Derived] Xie L, Sun X, Xu J, Liang X, Liu K, Sun K, Yang R, Tang X, Guo W. The efficacy and safety of vincristine, irinotecan and anlotinib in Epithelioid Sarcoma. BMC Cancer. 2024 Feb 3;24(1):172. doi: 10.1186/s12885-024-11921-7. PMID 38310286